CLINICAL TRIAL: NCT00598806
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind, Phase 3 Trial of Single-Dose Intravesical Apaziquone (EOquin®) as a Surgical Adjuvant Instilled in the Early Postoperative Period in Patients Undergoing Transurethral Resection for Noninvasive Bladder Cancer (Protocol SPI-612)
Brief Title: Single Dose Intravesical Apaziquone Postoperative in Patients Undergoing TURBT for Noninvasive Bladder Cancer (SPI-612)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-612
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Bladder Cancer
Keywords: Noninvasive Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — apaziquone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apaziquone (Experimental): TURBT + a single intravesical dose of Apaziquone 4mg in 40ml instilled into the bladder post-TURBT
  Interventions: Drug: Apaziquone; Procedure: TURBT
- Placebo (Placebo Comparator): TURBT + a single intravesical dose of placebo instilled into the bladder post-TURBT
  Interventions: Drug: Placebo; Procedure: TURBT

INTERVENTIONS:
Drug: Apaziquone — A single intravesical dose of Apaziquone 4mg in 40ml instilled into the bladder post-TURBT
  Other Names: EOquin®, Qapzola
  Arms: Apaziquone
Drug: Placebo — A single intravesical dose of placebo instilled into the bladder post-TURBT
  Arms: Placebo
Procedure: TURBT — TransUrethral Resection of the Bladder Tumor

SUMMARY:
The purpose of this study was to evaluate the 2-Year Recurrence Rate of bladder cancer in randomized patients with tumor histology Ta, G1-G2 who received TransUrethral Resection of Bladder Tumor (TURBT) plus apaziquone versus those who received TURBT plus placebo.

DETAILED DESCRIPTION:
This was a Phase 3, multicenter, randomized, double-blind, placebo-controlled study. Within 14 days of Screening, eligible patients underwent a TURBT during Visit 1 (Day 0) following which they were immediately randomized in a 1:1 ratio to receive either placebo or 4 mg apaziquone, instilled in a volume of 40 mL into the bladder within 6 hours from the end of the TURBT procedure. After a 60-minute retention period, study drug was drained from the bladder.

A postoperative follow-up examination and review of the local pathology report were performed at Visit 2, which occurred 21 days (±10 days) after the TURBT (Week 3).

* If the histology of the patient's tumor was confirmed as Ta, G1-G2 (ie, low grade according to World Health Organization [WHO]/International Society of Urologic Pathology [ISUP] classification), no further treatment was given and the patient was observed cystoscopically every 3 months through Year 2 for tumor recurrence (Visit 3 through Visit 10).
* If the histology of the patient's tumor was other than Ta, G1 or G2 (low grade [WHO/ISUP classification]), further treatment was given in accordance with current treatment guidelines, and the patient was followed up cystoscopically every 3 months through Year 2 for tumor recurrence (Visit 3 through Visit 10).

All patients were to be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

All of the following questions must be answered "Yes" in order for the patient to participate in the study.

1. Has the patient given written informed consent?
2. Is the patient at least 18 years old?
3. Does the patient have transitional cell carcinoma of the bladder with clinically apparent tumor Ta, grade G1-G2?
4. If the patient is a female of childbearing potential, is she using an acceptable/effective method of contraception?
5. If the patient is a female of childbearing potential, has she had a negative serum pregnancy test within the past 14 days?
6. Is the patient willing and able to abide by the protocol?

Exclusion Criteria:

All of the following questions must be answered "No" in order for the patient to participate in the study.

1. Does the patient have more than 5 bladder tumors?
2. Does any single bladder tumor exceed 3.5 cm in diameter?
3. Does the patient have a single, primary bladder tumor <0.5 cm and has no previous diagnosis of bladder cancer?
4. Has the patient ever received EOquin(r)?
5. Does the patient have, or has the patient ever had, any bladder tumor known to be other than tumor Ta or grade G1 or G2 (low grade [WHO/ISUP classification])?
6. Does the patient have, or has the patient ever had any bladder tumor with histology other than transitional cell carcinoma?
7. Does the patient have, or has the patient ever had, carcinoma in situ (CIS)?
8. Does the patient have an active urinary tract infection?
9. Does the patient have a bleeding disorder or a screening platelet count < 100 x 109/L?
10. Does the patient have any unstable medical condition that would make it unsafe for him/her to undergo TURBT under general or spinal anesthesia?
11. Does the patient have screening hemoglobin < 10 mg/dL, a screening absolute neutrophil count < 1.5 x 109/L?
12. Does the patient have a known immunodeficiency disorder?
13. Has the patient received any investigational treatment within the past 30 days?
14. Is the patient breast feeding?
15. Does the patient have a history of interstitial cystitis?
16. Does the patient have a history of allergy to red color food dye?
17. Has the patient had transitional cell carcinoma of the bladder within the past 4 months?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shanta Chawla, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (77):
- United States (21):
  - Advanced Urology Medical Center Clinical Trials, Anaheim, California
  - Hal J. Bashein, D.O., West Palm Beach, Florida
  - Urology Enterprises, Marietta, Georgia
  - North Fulton Urology, Roswell, Georgia
  - Hines VA Hospital, Hines, Illinois
  - The Urology Center, Slidell, Louisiana
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Towson, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - PharmaTrials, Inc. - Male & Female Urology, Hillsborough, New Jersey
  - PharmaTrials, Inc., Hillsborough, New Jersey
  - Medical & Clinical Research Associates, LLC, Bay Shore, New York
  - Urology Associates, PC, Manhasset, New York
  - North Shore - LIJ Health System - The Arthur Smith Institute for Urology, New Hyde Park, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Center for Urologic Care, Bryn Mawr, Pennsylvania
  - Medical University of South Carolina, Dept. of Urology, Charleston, South Carolina
  - Urology Associates of South Texas, McAllen, Texas
  - Salt Lake Research, Salt Lake City, Utah
  - Adult and Pediatric Urologists, Alexandria, Virginia
- Canada (32):
  - Prostate Cancer Institute, Calgary, Alberta
  - Lintor Medical, Inc., North Vancouver, British Columbia
  - Andreou Research, Surrey, British Columbia
  - Can-Med Clinical Research, Inc, Victoria, British Columbia
  - G. Steinhoff Clinical Research, Victoria, British Columbia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - The Male/Female Health and Research Center - Royal Court Medical Centre, Barrie, Ontario
  - Brantford Urology Research, Brantford, Ontario
  - G. Kenneth Jansz Medicine Professional Corporation, Burlington, Ontario
  - Urology Resource Centre, Burlington, Ontario
  - Kingston General Hospital / Queen's University, Kingston, Ontario
  - Urology Associates, Urologic Medical Research, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Mor Urology, Inc., Newmarket, Ontario
  - Dr. Bernard Goldfarb, North Bay, Ontario
  - Stanley Flax Medical Professional Corporation, North York, Ontario
  - The Fe/Male Health Centre, Oakville, Ontario
  - Orillia Urology Associates, Orillia, Ontario
  - Urotec, Oshawa, Ontario
  - ADA Medical Ltd., Peterborough, Ontario
  - AGT Research, Scarborough Village, Ontario
  - Urology & Male Infertility, Scarborough Village, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network Princess Margaret Hospital, Toronto, Ontario
  - The Male Health Centre, Toronto, Ontario
  - Saint Joseph Health Center, Toronto, Ontario
  - UroLaval, Laval, Quebec
  - McGill Urology Associates, Montreal, Quebec
  - Ultra-Med, Inc., Pointe Clare, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Centre hospitalier universitaire de Quebec, Québec
- Poland (24):
  - Uniwersytecki Szpital Kliniczny, Bialystok
  - Szpital Wojewódzki w Bielsku-Białej, Bielsko-Biala
  - Akademickie Centrum Kliniczne - Szpital Akademii Medycznej w Gdańsku, Gdansk
  - Publiczny Specjalistyczny Zakład Opieki Zdrowotnej w Inowrocławiu, Inowrocław
  - Szpital Miejski im. Prof. E. Michałowskiego, Katowice
  - Świętokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakład Opieki Zdrowotnej, Kielce
  - Szpital Specjalistyczny w Kościerzynie, Kościerzyna
  - Niepubliczny Zakład Opieki Zdrowotnej "Racławicka", Krakow
  - Uniwersytecki Szpital Kliniczny nr 2 Wojskowej Akademii Medycznej Uniwersytetu Medycznego w Łodzi - Centralny Szpital Weteranów, Lodz
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Lublin
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej w Pabianicach, Pabianice
  - Zakład Opieki Zdrowotnej Poznań - Stare Miasto, Poznan
  - Szpital Kolejowy im. Dr med.. Włodzimierza Roeflera w Pruszkowie, Pruszków
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej, Wojewódzki Szpital Specjalistyczny nr 3, Rybnik
  - Wojewódzki Szpital Specjalistyczny W Siedlcach, Siedlce
  - Pomorska Akademia Medyczna, Szczecin
  - Wojewódzki Szpital Specjalistyczny im Janusza Korczaka, Słupsk
  - Centrum Medycznego Kształcenia Podyplomowego, Samodzielny Publiczny Szpital Kliniczny im. Prof. W. Orłowskiego, Warsaw
  - Wojskowy Instytut Medyczny, Centralny Szpital Kliniczny MON, Warsaw
  - Szpital Kliniczny Dzieciątka Jezus - Centrum Leczenia Obrażeń, Warsaw
  - Centrum Onkologii im. Marii Skodowskiej-Curie, Warsaw
  - Fundacja "Urologia", Międzyleski Szpital Specjalistyczny w Warszawie, Warsaw
  - Akademicki Szpital Kliniczny im Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Ośrodek Badawczo Rozwojowy, Wroclaw

RESULTS

PARTICIPANT FLOW:
Groups:
- Apaziquone: Apaziquone: TURBT + a single intravesical dose of Apaziquone 4mg in 40ml instilled into the bladder post-TURBT
- Placebo: Placebo: TURBT + a single intravesical dose of placebo instilled into the bladder post-TURBT
Period: Overall Study
Arm/Group | Apaziquone | Placebo
Started | 402 | 410
Completed | 329 | 346
Not Completed | 73 | 64

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Apaziquone | Placebo | Total
Number analyzed (Participants) | 402 | 410 | 812
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (11.60) | 66.5 (11.83) | 66.7 (11.71)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 157 | 164 | 321
  65-75 | 144 | 146 | 290
  >75 | 101 | 100 | 201
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 108 | 213
  Male | 297 | 302 | 599
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 389 | 398 | 787
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 392 | 400 | 792
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 215 | 223 | 438
  United States | 82 | 85 | 167
  Poland | 105 | 102 | 207

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Rate at 2 Years
Description: The percentage of participants with histologically confirmed recurrence of the bladder tumor at any time after randomization and on or before year 2.
Time Frame: 2 years
Population: Target Ta, G1-G2 Population: patients who had 4 or fewer tumors that were ≤ 3.5 cm each at the time of randomization and who had subsequent histological confirmation from the central pathology lab that the tumors resected at the time of randomization were Ta, Grade 1 or 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 282 | 298
Participants
  Recurrence | 112 | 138
  Non-Recurrence | 170 | 160
Statistical Analysis 1: Comparison: Apaziquone vs Placebo; Test type: Superiority; p = 0.1094, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.55 to 1.06]

2. Secondary Outcome: Time to Recurrence
Description: The number of months from randomization to histologically confirmed recurrence of the patient's bladder tumor.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 282 | 298
months | 18.1 (0.5) | 16.7 (0.5)
Statistical Analysis 1: Comparison: Apaziquone vs Placebo; Test type: Superiority; p = 0.1038, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.63 to 1.04]

3. Secondary Outcome: Progression Rate at 2 Years
Description: The percentage of participants that progress to either a higher stage or grade from the histologically confirmed stage and grade at time of randomization.
Time Frame: 2 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 282 | 298
Participants
  Progression | 29 | 37
  Non-Progression | 253 | 261

4. Secondary Outcome: Time to Progression
Description: The number of months from randomization to progression to either a higher stage or grade of the patient's bladder tumor.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 282 | 298
months | 22.7 (0.3) | 21.9 (0.29)

5. Secondary Outcome: Number of Recurrences Per Patient
Description: The number of histologically confirmed recurrences during the course of the study.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: recurrences
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 282 | 298
recurrences | 0.6 (0.98) | 0.9 (1.19)

6. Secondary Outcome: Disease-Free Interval
Description: The number of months from randomization to histologically confirmed progression of the patient's bladder tumor or death from any cause
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 282 | 298
months | 22.7 (0.3) | 21.9 (0.29)

7. Secondary Outcome: Disease-Free Survival
Description: The number of months from randomization to histologically confirmed recurrence of the patient's bladder tumor or death from any cause
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 282 | 298
months | 17.9 (0.5) | 16.4 (0.5)

8. Secondary Outcome: Overall Survival
Description: The number of months from randomization to death from any cause.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 282 | 298
months | 24 (0.14) | 20.2 (0.12)

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (ie, AEs that occurred or worsened following the TURBT procedure) were recorded from the time of randomization to Month 6; after Month 6 until Month 24 (end of study), only genitourinary AEs and Serious AEs (SAEs) were recorded.
Groups:
- Apaziquone: Apaziquone: TURBT + a single intravesical dose of EOquin® 4mg in 40ml instilled into the bladder post-TURBT
Arm/Group | Apaziquone | Placebo
All-Cause Mortality (participants affected / at risk) | 14/402 | 14/410
Serious Adverse Events (participants affected / at risk) | 96/402 | 108/410
Other Adverse Events (participants affected / at risk) | 313/402 | 322/410
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apaziquone (N=402) | Placebo (N=410)
Urinary retention (Renal and urinary disorders) | 8 | 4
Cardiac failure congestive (Cardiac disorders) | 7 | 1
Hematuria (Renal and urinary disorders) | 5 | 12
Cerebrovascular accident (Nervous system disorders) | 4 | 5
Renal failure acute (Renal and urinary disorders) | 4 | 2
Hydronephrosis (Renal and urinary disorders) | 4 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Knee arthroplasty (Surgical and medical procedures) | 3 | 4
Pneumonia (Infections and infestations) | 3 | 3
Transurethral prostatectomy (Surgical and medical procedures) | 3 | 2
Bladder perforation (Renal and urinary disorders) | 3 | 1
Hip arthroplasty (Surgical and medical procedures) | 2 | 4
Urinary bladder hemorrhage (Renal and urinary disorders) | 2 | 3
Cardiac arrest (Cardiac disorders) | 2 | 2
Coronary artery disease (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 2 | 2
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 2 | 2
Cardiogenic shock (Cardiac disorders) | 2 | 1
Urosepsis (Infections and infestations) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Ureteric obstruction (Renal and urinary disorders) | 2 | 0
Aortic aneurysm repair (Surgical and medical procedures) | 2 | 0
Radiotherapy (Surgical and medical procedures) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Radical prostatectomy (Surgical and medical procedures) | 1 | 2
Angina unstable (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 1
Death (General disorders) | 1 | 1
Post procedural hematuria (Injury, poisoning and procedural complications) | 1 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chest pain (General disorders) | 0 | 3
Angina pectoris (Cardiac disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Enterovesical fistula (Gastrointestinal disorders) | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 2
Cystocele repair (Surgical and medical procedures) | 0 | 2
Circulatory collapse (Vascular disorders) | 0 | 2
Femoral artery occlusion (Vascular disorders) | 0 | 2
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Implant site erosion (General disorders) | 1 | 0
Infusion site thrombosis (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Hypovolemia (Metabolism and nutrition disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 1 | 0
Transient ischemic attack (Nervous system disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Bladder neck obstruction (Renal and urinary disorders) | 1 | 0
Urethral hemorrhage (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arterial aneurysm repair (Surgical and medical procedures) | 1 | 0
Arteriovenous graft (Surgical and medical procedures) | 1 | 0
Carotid endarterectomy (Surgical and medical procedures) | 1 | 0
Coronary angioplasty (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair (Surgical and medical procedures) | 1 | 0
Urethral operation (Surgical and medical procedures) | 1 | 0
Urethrotomy (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Leriche syndrome (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Intestinal strangulation (Gastrointestinal disorders) | 0 | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Ascariasis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Catheterisation cardiac (Investigations) | 0 | 1
Urine cytology abnormal (Investigations) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral hemorrhage (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bladder irrigation (Surgical and medical procedures) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Hemorrhoid operation (Surgical and medical procedures) | 0 | 1
Nephrectomy (Surgical and medical procedures) | 0 | 1
Prostatectomy (Surgical and medical procedures) | 0 | 1
Radical mastectomy (Surgical and medical procedures) | 0 | 1
Spinal decompression (Surgical and medical procedures) | 0 | 1
Ureteric calculus removal (Surgical and medical procedures) | 0 | 1
Urinary cystectomy (Surgical and medical procedures) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apaziquone (N=402) | Placebo (N=410)
Urinary tract infection (Infections and infestations) | 87 | 90
Procedural pain (Injury, poisoning and procedural complications) | 14 | 21
Bladder pain (Renal and urinary disorders) | 30 | 25
Dysuria (Renal and urinary disorders) | 86 | 62
Haematuria (Renal and urinary disorders) | 69 | 73
Micturition urgency (Renal and urinary disorders) | 31 | 37
Pollakiuria (Renal and urinary disorders) | 43 | 39
Urinary retention (Renal and urinary disorders) | 26 | 26
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 17 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
First publication is the multi-center publication of Study results from all study sites. Other than the multi-center publication, site may publish an independent publication of data generated by site subject to Sponsor review rights (e.g., review for intellectual property, confidentiality).